CLINICAL TRIAL: NCT03415984
Title: Evaluation of the Prevalence of Age Related Macular Degeneration (ARMD) in Parkinson's Patients and Assesment of the Role of L-DOPA (AMD-PARK)
Brief Title: Prevalence of Age Related Macular Degeneration (ARMD) in Parkinson's Patients and Assesment of the Role of L-DOPA
Acronym: AMD-PARK
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMT_2017_24
Record Dates: First submitted 2018-01-19; First posted 2018-01-30 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease; Age Related Macular Degeneration
Keywords: Parkinson Disease; Age Related Macular Degeneration; L-DOPA
MeSH Terms: conditions — Parkinson Disease; Macular Degeneration | interventions — Tomography, Optical Coherence; Optical Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed patients: Patients with Parkinson's disease treated with L-DOPA
  Interventions: Diagnostic Test: Color retinography; Diagnostic Test: Optical coherence tomography; Diagnostic Test: Fundus autofluorescence imaging
- Non exposed patients: Patients with Parkinson's disease not treated with L-DOPA
  Interventions: Diagnostic Test: Color retinography; Diagnostic Test: Optical coherence tomography; Diagnostic Test: Fundus autofluorescence imaging

INTERVENTIONS:
Diagnostic Test: Color retinography — Color retinography
Diagnostic Test: Optical coherence tomography — Optical coherence tomography
Diagnostic Test: Fundus autofluorescence imaging — Fundus autofluorescence imaging

SUMMARY:
Age related macular degeneration (ARMD) is a major and irreversible cause of blindness among the elderly. The sub-retinal space, located between the retinal pigmentary epithelium (RPE) and the external segments of the retinal photoreceptors, plays a crucial role in this pathology. A recent epidemiologic study in the US, has shown that Parkinson patients treated with L-DOPA, developed only later an ARMD when compared to the untreated patients.

The L-Dopa is an endogenous ligand of the GPR43 receptor (G protein-coupled receptors), located on the RPE's cell's apical pole.

This receptor, via several intracellular mechanisms, regulates the cell's exosomal and endosomal pathways: it would appear that the L-DOPA, by stimulating this receptor, decreases significantly the RPE's exosome release.

The contents of the exosomes is still uncertain, however in addition to their signalization role, it seems they transport pro-inflammatory components, possibly helping the cellular recruitment due to the mononuclear phagocytic systems, particularly toxic for the photoreceptors.

The aim of this study is to estimate the prevalence of ARMD in a sample of Parkinson's Patients followed at Fondation Ophtalmologique Adolphe de Rothschild and to compared it to the prevalence of ARMD of the general population.

Furthermore the study aims to explore a possible causal link between L-DOPA treatment and ARMD.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged of 50 years old and more
* Parkinson's disease

Exclusion Criteria:

* Patient under a measure of legal protection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease, treated or not treated with L-DOPA
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of ARMD | baseline
  Comparison of the percentage of patients with ARMD in both groups (Parkinson's Patients treated or not treated with L-DOPA) : Diagnosis of ARMD by the ophthalmologist is based on 3 exams (Color retinography, Optical coherence tomography and Fundus autofluorescence imaging). In case of any discrepancy between the results of the 3 exams, the final diagnosis of ARMD is based on the Optical coherence tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Martine MAUGET FAYSSE, MD, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation ophtalmologique Adolphe de Rothschild, Paris, France